CLINICAL TRIAL: NCT02537522
Title: Evaluation of 8.5 vs 9.0 Base Curve for 1-DAY ACUVUE(r) TruEye(r) Brand Contact Lenses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CR-5730
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Contact Lens Base Curve (BC) Fit and Comfort
MeSH Terms: interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Test/Control - Phase 1 (Experimental): Over visits 1 and 2, subject will wear Contact Lenses with 8.5 BC in right eye and Contact Lenses with 9.0 BC in left eye in a contralateral manner.
  Interventions: Device: Contact Lenses with 8.5 BC; Device: Contact Lenses with 9.0 BC
- Control/Test - Phase 1 (Experimental): Over visits 1 and 2, subject will wear Contact Lenses with 9.0 BC in right eye and Contact Lenses with 8.5 BC in left eye in a contralateral manner.
  Interventions: Device: Contact Lenses with 8.5 BC; Device: Contact Lenses with 9.0 BC
- Test/Control - Phase 2 (Experimental): During Phase 2, subjects will wear a pair of Contact Lenses with 9.0 BC at Period 1 and Contact Lenses with 8.5 BC at Period 2 in a bilateral manner.
  Interventions: Device: Contact Lenses with 8.5 BC; Device: Contact Lenses with 9.0 BC
- Control/Test - Phase 2 (Experimental): During Phase 2, subjects will wear a pair of Contact Lenses with 8.5 BC at Period 1 and Contact Lenses with 9.0 BC at Period 2 in a bilateral manner.
  Interventions: Device: Contact Lenses with 8.5 BC; Device: Contact Lenses with 9.0 BC

INTERVENTIONS:
Device: Contact Lenses with 8.5 BC — Subjects will wear the marketed, daily disposable contact lenses in 8.5 BC.
  Other Names: Marketed Daily Disposable Soft Contact Lenses
Device: Contact Lenses with 9.0 BC — Subjects will wear the marketed, daily disposable contact lenses in 9.0 BC.
  Other Names: Marketed Daily Disposable Soft Contact Lenses

SUMMARY:
The objective of this study is to determine if corneal diameter and keratometry readings correlate to subjective comfort and lens fitting characteristics.

ELIGIBILITY:
Inclusion Criteria:

* The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
* The subject must be no less than 18 and no more than 45 years of age with no presbyopic add.
* The subject must be willing and able to adhere to the instructions set out in the protocol.
* The subject must be an adapted soft contact lens wearer in both eyes.
* The subject must be willing to wear the study contact lenses up to 14 hours/day.
* The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 Diopters (D) to -6.00 D in each eye.
* The subject must have refractive cylinder less than or equal to 1.00 D in each eye.
* The subject must have best corrected visual acuity of 20/30 (6/9) or better in each eye.
* The subject must require a visual correction in both eyes (no monofit or monovision allowed).
* The subject must have normal eyes (i.e., no ocular medications or infections of any type).

Exclusion Criteria:

* Current 1-DAY ACUVUE® TruEye® wearers
* Anisometropia of 1.00 D or greater
* Any Ocular or systemic allergies or diseases which might interfere with contact lens wear.
* Any Systemic disease, autoimmune disease, or use of medication which might interfere with contact lens wear.
* Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
* Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
* Any ocular infection
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear
* Pregnancy or lactation
* Diabetes
* Infectious diseases (e.g. hepatitis, tuberculosis) or an immuno-suppressive disease (e.g. HIV).
* Employee of investigational clinic (e.g., Investigator, Coordinator, Technician)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 72 subjects were enrolled into this study. Of the enrolled subjects 1 did not meet the eligibility criteria and 71 were dispensed lenses. Of the dispensed subjects 45 completed both Phase I and II while 26 subjects were discontinued.
Groups:
- Test/Control - Phase 1: Subjects randomized to this sequence in Phase I wore the test lens narafilcon A with 8.5 Base Curve in their left eye and then wore the narafilcon A with 9.0 Base Curve in their right eye.
- Control/Test - Phase 1: Subjects randomized to this sequence in Phase I wore the test lens narafilcon A with 9.0 Base Curve in their left eye and then wore the narafilcon A with 8.5 Base Curve in their right eye.
- Test/Control - Phase 2: Subjects randomized to this sequence in Phase II wore the narafilcon A lens with 8.5 Base Curve in both eyes and then wore narafilcon A lens with 9.0 Base Curve in both eyes.
- Control/Test - Phase 2: Subjects randomized to this sequence in Phase II wore the narafilcon A lens with 9.0 Base Curve in both eyes and then wore narafilcon A lens with 8.5 Base Curve in both eyes.
Period: Phase I - Contralateral
Arm/Group | Test/Control - Phase 1 | Control/Test - Phase 1 | Test/Control - Phase 2 | Control/Test - Phase 2
Started | 34 | 37 | 0 | 0
Completed | 19 | 27 | 0 | 0
Not Completed | 15 | 10 | 0 | 0
Not completed — Subject no longer eligible | 15 | 7 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — incorrect randomization | 0 | 1 | 0 | 0
Not completed — unsatisfactory lens fitting | 0 | 1 | 0 | 0
Period: Phase II - Period 1 Bilateral
Arm/Group | Test/Control - Phase 1 | Control/Test - Phase 1 | Test/Control - Phase 2 | Control/Test - Phase 2
Started | 0 | 0 | 23 | 23
Completed | 0 | 0 | 23 | 22
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Phase II - Period 2 Bilateral
Arm/Group | Test/Control - Phase 1 | Control/Test - Phase 1 | Test/Control - Phase 2 | Control/Test - Phase 2
Started | 0 | 0 | 23 | 22
Completed | 0 | 0 | 23 | 22
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed at least one study lens.
Groups:
- Dispensed Subjects: All subjects that were dispensed at least one study lens throughout the course of the study.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Subjective CLUE Comfort and Keratometry
Description: CLUE- The Contact Lens User Evaluation (CLUE)™ questionnaire is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20) with a range of 0-120, where higher scores indicate a more favorable/positive response (Wirth, RJ. Et al. August 2016). Keratometry measurements of major keratometric meridians (diopter [DK]) and their location (degrees) was collected at baseline for both eyes. The correlation between CLUE comfort and maximum Keratometry measurements of the two eyes within each subject and the correlation between CLUE comfort and the minimum Keratometry measurements of the two eyes within each subject were reported.
Time Frame: 3-day follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Pearson Correlation
Groups:
- Narafilcon A- 8.5 Base Curve: Subjects that wore the narafilcon A lens with 8.5 Base Curve in either the 1st or 2nd period of the study during either Phase II.
- Narafilcon A- 9.0 Base Curve: Subjects that wore the narafilcon A lens with 9.0 Base Curve in either the 1st or 2nd period of the study during either Phase II.
Arm/Group | Narafilcon A- 8.5 Base Curve | Narafilcon A- 9.0 Base Curve
Number analyzed (Participants) | 43 | 43
Pearson Correlation
  Minimum Keratometry measurements | 0.042 | 0.004
  Maximum Keratometry measurements | -0.001 | -0.002

2. Primary Outcome: Correlation Between Subjective CLUE Comfort and Corneal Diameter
Description: Assessment The Contact Lens User Evaluation (CLUE)™ questionnaire is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20) with a range of 0-120, where higher scores indicate a more favorable/positive response (Wirth, RJ Et al. August 2016). Corneal diameter (horizontal visible iris diameter [HVID]) was collected at baseline for both eyes using a slit lamp reticle, measuring to the nearest 0.05 mm.The maximum (or minimum) measurements of HVID between the two eyes of each subject were used for correlation analyses between subjective CLUE comfort score and corneal diameter.
Time Frame: 3-day follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Pearson Correlation
Arm/Group | Narafilcon A- 8.5 Base Curve | Narafilcon A- 9.0 Base Curve
Number analyzed (Participants) | 43 | 43
Pearson Correlation
  Minimum Corneal diameter | 0.011 | -0.086
  Maximum Corneal diameter | 0.021 | -0.119

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 1-week per subject.
Arm/Group | Narafilcon A- 8.5 Base Curve | Narafilcon A- 9.0 Base Curve
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71
Other Adverse Events (participants affected / at risk) | 0/71 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days